CLINICAL TRIAL: NCT02704728
Title: A Randomised, Double-blind, Placebo-controlled Study to Assess the Safety and Tolerability of Bacteroides Thetaiotaomicron in Young People Aged 16 to 18 Years With Stable Crohn's Disease
Brief Title: Study of Bacteroides Thetaiotaomicron in Young People Aged 16 to 18 Years With Stable Crohn's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: 4D pharma plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Theta 001
Record Dates: First submitted 2016-01-12; First posted 2016-03-10 (Estimated); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Thetanix (Experimental): In Part A, 8 subjects will receive a single dose and in Part B, 8 subjects will receive twice daily doses for 7.5 days (a total of 15 doses). Each dose consists of three capsules
  Interventions: Other: Thetanix
- Placebo (Placebo Comparator): In Part A, 2 subjects will receive a single dose and in Part B, 2 subjects will receive twice daily doses for 7.5 days (a total of 15 doses). Each dose consists of three capsules.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Thetanix — Thetanix is an encapsulated lyophilised formulation of a pure culture of Bacteroides thetaiotaomicron with excipients.
  Other Names: B. theta
  Arms: Thetanix
Other: Placebo — Placebo is encapsulated microcrystalline cellulose without Bacteroides thetaiotaomicron.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety and tolerability of Bacteroides thetaiotaomicron (Thetanix®)) capsules in young people aged 16 to 18 years with stable Crohn's disease.

DETAILED DESCRIPTION:
This study is a single (Part A) and multiple (Part B) dose study. Following informed consent and screening, 10 eligible subjects will receive a single dose of Thetanix or placebo in the clinic. A Safety Review Committee will review the safety data up to Day 7 from these first ten subjects and determine if it is appropriate to continue into Part B in which 10 subjects will receive 15 doses of Thetanix or placebo in a twice daily dosing regimen over 7.5 days. In both parts of the study, 8 of the 10 subjects will randomly receive Thetanix and 2 subjects will randomly receive placebo. Each dose consists of three capsules. Subjects in Part B will receive the first and last dose in the clinic and will take 13 doses at home. While at home, subjects will be required to answer questions about their health, record their body temperature and when they take the capsules in an electronic diary. Subjects developing a fever will undergo further assessments, including blood cultures. Subjects will provide stool samples for analysis of microbiota and faecal calprotectin.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 16 to 18 years inclusive, with confirmed diagnosis of Crohn's disease who are currently in clinical remission* in the opinion of the investigator and who are otherwise healthy.
2. Subjects who are able and willing to give written informed consent to participate. If applicable, a parent/carer may also give consent to their participation.

Exclusion Criteria:

1. Subjects who are pregnant or breastfeeding.
2. Subject who are experiencing an exacerbation at the time of screening or up to the time of the first dose.
3. Subjects who have undergone previous surgery for resection of bowel.
4. Subjects who have fistulisation.
5. Subjects who have had a significant change in their immune-modulating maintenance medication in the 3 months prior to screening and/or the start of dosing.
6. Subjects who have taken systemic steroids in the last 3 months.
7. Subjects who are unable to take any oral feeding.
8. Subjects with feeding gastrostomies.
9. Subjects who have non-food dietary supplementation for any reason changed within 1 month prior to dosing.
10. Subjects who have received monoclonal antibodies in the 6 months prior to dosing.
11. Subjects who have received antibiotics or probiotic dietary supplementation in the two weeks before dosing. Subjects who have received foods with probiotics e.g. yoghurts will be permitted to volunteer for the study.
12. Subjects who are receiving exclusive enteral feeding or have completed a course of exclusive enteral feeding in the 3 months prior to dosing.
13. Subjects with concomitant autoimmune diseases.
14. Female Subjects of child bearing potential unwilling to use effective contraception from the signing of the consent form until completion of two periods after the last dose. An effective method of birth control is defined as one which results in a low failure rate (i.e. less than 1% per year) when used consistently and correctly such as sterilisation, implants, injectables, combined oral contraceptives, Intrauterine Device (IUD), condoms, occlusive caps (cervical/vault caps) with spermicidal foam/gel/film/cream/pessary. True sexual abstinence is acceptable when this is in line with the preferred and usual lifestyle of the subject.
15. Subjects with clinically significantly, in the opinion of the investigator, elevated platelets, white cell count, C-reactive protein, erythrocyte sedimentation rate (ESR), low albumin or haemoglobin.
16. Subjects who are positive for the following viruses: HIV, hepatitis B and hepatitis C.
17. Subjects who smoke cigarettes or use other tobacco or nicotine containing products, including e-cigarettes.
18. Subjects who have a known sensitivity to any of the constituents of the investigational medicinal compound.
19. Diastolic blood pressure <50 or >90 mmHg, a systolic blood pressure <100 or >150 mmHg, a pulse <40 or >100 beats per minute (bpm) after resting for 5 minutes.
20. Subjects with clinically significantly abnormal ECGs or structural cardiac abnormalities e.g. valvular heart disease, patent foramen ovale.
21. BMI Z SCORE less than -2.6 or greater than 2.6 (0 ± 2.6); i.e. below the 2nd centile or greater than the 98th centile.
22. Any condition that, in the opinion of the Investigator, might interfere with the primary study objective.
23. Subjects allergic to metronidazole and co-amoxiclav

Ages: 16 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events | Part A (single dose): Day 7. Part B (15 doses over 7.5 days): Day 14
  The change from baseline will be assessed at Day 7 (Part A) and at Day 14 (Part B). Part A and Part B will be analysed separately as they are of different duration. The primary endpoint for each part is taken as 7 days after the last dose.

SECONDARY OUTCOMES:
Physician Global Assessment | Part B: Day 14
  Change in Physician Global Assessment
Weighted Paediatric Crohn's Disease Activity Index | Part B; Day 14
  Change in Weighted Paediatric Disease Activity Index
The number of subjects with abnormal clinically and non-clinically significant or out of expected range tests. | Part A: Day 7; Part B: Day 14
  Tests include: Serum biochemistry and haematology; physical examinations, blood pressure, pulse rate, respiratory rate and oral temperature, weight, height, ECG parameters.
Part A: Faecal Microbiome Part B Microbiome and faecal calprotectin concentrations | Part B: Day 14
  Stool samples will be collected and analysed for faecal calprotectin and microbial communities with specific interest in B. theta.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Hansen, MB ChB PhD FRCPCH, Principal Investigator — South Glasgow University Hospitals NHS Trust; David Wilson, MD DCH FRCP(Edin) FRCPCH, Principal Investigator — Royal Hospital for Sick Children Edinburgh
Locations (5):
- United Kingdom (5):
  - Birmingham Children's Hospital, Birmingham, Birmimgham
  - Clinical Research Facility, Edinburgh
  - Clinical Research Faciity, Glasgow
  - Alder Hey Children's Hospital, Liverpool
  - Barts Health NHS Trust, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hansen R, Sanderson IR, Muhammed R, Allen S, Tzivinikos C, Henderson P, Gervais L, Jeffery IB, Mullins DP, O'Herlihy EA, Weinberg JD, Kitson G, Russell RK, Wilson DC. A Double-Blind, Placebo-Controlled Trial to Assess Safety and Tolerability of (Thetanix) Bacteroides thetaiotaomicron in Adolescent Crohn's Disease. Clin Transl Gastroenterol. 2020 Dec 18;12(1):e00287. doi: 10.14309/ctg.0000000000000287. PMID 33464732